CLINICAL TRIAL: NCT07360158
Title: Post-market Study for the CorSky Family of ICDs
Brief Title: BIO|MASTER.CorSky Family Post-market Study for the CorSky Family of ICDs
Status: Not yet recruiting | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: TA121
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Tachycardia, Heart Failure
MeSH Terms: conditions — Tachycardia; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CorSky ICD or CRT-D — Subjects with an indication for an ICD or CRT-D device will be implanted with a CorSky device of the CorSky ICD family according to standard implantation procedures. Device programming will be done according to the medical needs of the subjects.

SUMMARY:
The CorSky family is BIOTRONIK´s new generation of ICDs. They are the successor devices of the current Acticor/Rivacor family and inherit all iShock/iShock_BC (Ilivia Neo, Intica Neo) implant and programmer software features.

The new features of CorSky Family are either true novel BIOTRONIK ICD features or mainly driven by unification with the Amvia pacemaker family (Amvia Edge, -Sky).

The goal of the study is to confirm the safety and performance of the CorSky Family of ICDs and CRT-Ds.

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for ICD or CRT-D therapy according to clinical guidelines
* Planned for de novo implantation of an ICD/CRT-D, or upgrade/exchange from existing ICD/CRT-D or pacemaker
* Ability to understand the nature of the study.
* Ability and willingness to perform all on-site follow-up visits at the study site.
* Ability and willingness to use the CardioMessenger and acceptance of the BIOTRONIK Home Monitoring® concept.

Exclusion Criteria:

* For VR-T DX and CRT-DX: Permanent atrial tachyarrhythmia
* For VR-T DX and CRT-DX: Patients requiring atrial pacing
* Planned for His-Bundle-Pacing
* Planned cardiac surgical procedures or interventional measures other than the study procedure within the next 12 months
* Pregnant or breast feeding.
* Age less than 18 years.
* Participation in an interventional clinical investigation in parallel to this study. ,
* Life-expectancy less than 12 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Standard indication for ICD or CRT-D
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
CorSky-related SADE-d free rate at 6 months | 6 months